CLINICAL TRIAL: NCT07146347
Title: A Trial to Evaluate Pharmacodynamics, Pharmacokinetics, Safety, and Tolerability of Insulin GZR4 Compared With Insulin Degludec and Insulin Icodec in Participants With Type 2 Diabetes
Brief Title: Comparison Study of Insulin GZR4 With Insulin Degludec
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GL-ULI-1001
Record Dates: First submitted 2025-08-18; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec; insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants will receive all three treatments in a fixed-sequence design. (Experimental): Each participant will undergo 3 treatment periods in a fixed-sequence design. In treatment Period 1, participants will receive insulin degludec once-daily for 7 days.
  In treatment Period 2, participants will receive GZR4, in treatment Period 3, participants will receive insulin icodec. Both GZR4 insulin and insulin icodec will be given once weekly over 6 weeks during two treatment periods.
  Interventions: Drug: GZR4 injection

INTERVENTIONS:
Drug: GZR4 injection — GZR4 is a new ultra-long-acting insulin analog
  Other Names: Degludec; Icodec

SUMMARY:
In this study, the investigational product will be compared with insulin degludec (Tresiba®) and insulin icodec (Awiqli®). The comparator products are approved for the treatment of T2DM in the European Union.

DETAILED DESCRIPTION:
This trial intends to investigate the pharmacodynamics, pharmacokinetics, safety, and tolerability of insulin GZR4 (hereafter referred to as GZR4) and estimate its potency in comparison with insulin degludec.

ELIGIBILITY:
Inclusion Criteria:

Signed and dated informed consent obtained before any trial-related activities. Trial-related activities are any procedures that would not have been done during normal management of the participant. 2. Male or female person with type 2 diabetes mellitus. 3. Age between 18 and 70 years, both inclusive. 4. Body Mass Index (BMI) between 27.0 and 38.0 kg/m^2, both inclusive. 5. Diabetes duration of at least 12 months. 6. Stable basal insulin regimen for at least 3 months. 7. Total daily basal insulin dose between 0.2-0.7 (I)U/kg/day, both inclusive. 8. HbA1c <= 9.0%. 9. Have venous access sufficient to allow cannulation for blood sampling as required by the protocol.

Exclusion Criteria:

Known or suspected hypersensitivity to IMPs or any of the excipients or to any component of the IMP formulations. 2. Previous participation in this trial. Participation is defined as randomized at Visit 2.

3. Receipt of any medicinal product in clinical development within 30 days or at least 5 half-lives of the related substances and their metabolites (whichever is longer) before randomization in this trial. 4. Use of insulin icodec as basal insulin. 5. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction. 6. Any history or presence of cancer except basal cell skin cancer or squamous cell skin cancer as judged by the investigator during the last 5 years prior to screening. 7. Clinically relevant comorbidity, capable of constituting a risk for the participant when participating in the trial or of interfering with the interpretation of data. Signs of acute illness as judged by the investigator. 9. Any serious systemic infectious disease during four weeks before randomization in this trial, as judged by the investigator. 10. Clinically significant abnormal values for hematology, biochemistry, coagulation, or urinalysis as judged by the investigator. 11. Estimated glomerular filtration rate (eGFR) < 60.0 mL/min/1.73m2. 12. Systolic blood pressure < 90 mmHg or >159 mmHg and/or diastolic blood pressure < 50 mmHg or > 99 mmHg at screening (one repeat test will be acceptable in case of suspected white-coat hypertension). 13. Heart rate at rest (as measured in vital sign assessment at screening) outside the range of 50-90 beats per minute at screening. This exclusion criterion also applies to participants who are on anti-hypertensives. 14. Clinically significant abnormal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in a supine position at screening, as judged by the investigator. 15. Proliferative retinopathy or maculopathy as judged by the investigator based on a recent (<1.5 years) ophthalmologic examination. 16. Severe neuropathy, in particular autonomic neuropathy, as judged by the investigator.

17. Recurrent severe hypoglycemia (more than 1 severe hypoglycemic episode requiring assistance from another person within 180 days before screening). 18. Hypoglycemic unawareness as judged by the investigator. 19. Hospitalization for diabetic ketoacidosis during the previous 6 months. 20. Use of oral antidiabetic drugs (OADs) within 1 month or 5 half-times (whichever is longer) prior to screening with the exception of stable doses (for at least 3 months prior to screening) of metformin, DPP4, SGLT2 inhibitors and GLP-1 receptor agonists. 21. Increased risk of thrombosis, e.g. participants with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the investigator. 22. Significant history of alcoholism or drug abuse as judged by the investigator or consuming more than 24.0 grams alcohol/day (for males), 12.0 grams alcohol/day (for females) on average. 23. A positive result in the alcohol and/or urine drug screen at the screening visit.

24. Smoking more than 5 cigarettes or the equivalent per day. 25. Inability or unwillingness to refrain from smoking and use of nicotine substitute products during the inpatient period Tested positive for hepatitis Bs antigen. 27. Tested positive for hepatitis C antibodies. (Presence of hepatitis C antibodies will not lead to exclusion if liver function tests are normal, and a hepatitis C polymerase chain reaction is negative). 28. Positive result to the test for HIV-1/2 antibodies or HIV-1 antigen. 29. Current treatment with systemically effective corticosteroids, monoamine oxidase inhibitors, systemic non-selective beta-blockers, growth hormone, non-routine vitamins or herbal products. 30. Use of non-prescription medication, including herbal products and non-routine vitamins, within 2 weeks prior screening that will interfere with PK of GZR4, insulin degludec or insulin icodec, as judged by the investigator. 31. Blood donation or blood loss of more than 500 mL within the last 3 months before screening.

32. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation. 33. Committed to an institution by virtue of an order issued either by the judicial or the administrative authorities. 34. If female, pregnancy or breast-feeding. 35. Women of childbearing potential who are not using a highly effective contraceptive method.

36. Men with non-pregnant partner(s) of childbearing potential not willing to use male contraception (condom) in addition to a highly effective contraceptive method during trial participation. 37. The investigator considers a person as unsuitable for inclusion in the trial for any other reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the PD of GZR4 compared to insulin degludec at steady state | 0 - 24 hours for Degulec 0-168 hours for GZR4
  AUCGIR.0-24h.ss, area under the glucose infusion rate curve over one dosing interval from 0 to 24 hours at steady state for insulin degludec
  AUCGIR.0-168h.ss, area under the glucose infusion rate curve over one dosing interval from 0 to 168 hours at steady state for GZR4

CONTACTS AND LOCATIONS:
Locations (1):
- Profil, Neuss, Germany